CLINICAL TRIAL: NCT06853301
Title: Towards a Smart Blood Culture Bottle: Machine Learning Assisted Electrochemical Profiling to Provide Early In-situ Identification of Bloodstream Infections Pathogens
Brief Title: Machine Learning Assisted Electrochemical Profiling to Provide Early Identification of Bloodstream Infections Pathogens
Acronym: E-MOC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: CEA - Leti (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 38RC24.0111_EMOC; 2024-A02517-40 (Other: ID RCB)
Record Dates: First submitted 2025-02-11; First posted 2025-02-28 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-02

CONDITIONS: Bacteremia Sepsis
Keywords: Rapid identification; Positive blood culture; Electrochemical profiling; Machine learning; Artificial intelligence; Bacteremia; Database
MeSH Terms: conditions — Bacteremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients (Experimental): Patients with blood culture sampling as standard of care. Two to four additional blood culture bottles sampled
  Interventions: Other: Blood culture sampling

INTERVENTIONS:
Other: Blood culture sampling — Patients with blood culture sampling as standard of care. Two to four additional blood culture bottles sampled that will be spiked with known bacterial species to determine their electrochemical profiles

SUMMARY:
In the context of a bacteremia, although significant progress has been made in speeding up pathogen identification once a blood culture bottle turns positive, few cost-effective solutions have been proposed to improve the earlier stages of the process-specifically, from blood collection to bottle positivity. The investigators propose that transport time could be leveraged to grow and identify bacteria, enabling faster access to actionable results through innovative technologies. This project aims to develop a bacterial identification database by analyzing the electrochemical profile of bacteria growing within the blood culture bottle, using machine learning.

ELIGIBILITY:
Inclusion Criteria:

* patient requiring a blood culture sample as standard of care procedure
* body weight > 50 Kg
* Patient for whom the collection of 2 to 4 additional blood culture bottles is feasible, depending on venous access
* patient who has not objected to participation in the project

Exclusion Criteria:

* Patient protected under the French Public Health Code (pregnant or breastfeeding women, patients under guardianship or curatorship, hospitalized under constraint, or deprived of liberty)
* patients with ongoing antibiotic treatment at the time of sampling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
List of samples with an electrochemical profile | From enrollment until the end of measurment of an electrochemical fingerprint in the blood cultures from the patient spiked with bacterial strains, assessed within up to one week after blood culture sampling
  List of samples (bacterial strain and corresponding pseudonymized blood culture) for which an electrochemical profile of the growing bacteria within the blood culture bottle was successfully obtained

SECONDARY OUTCOMES:
Identification performance | End of the study (18 months)
  Identification performance of electrochemical profiling of the growing bacteria followed by machine learning analysis

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Grenoble University Hospital, Grenoble
  - Hôpital AVICENNE (AP-HP), Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lamy B, Sundqvist M, Idelevich EA; ESCMID Study Group for Bloodstream Infections, Endocarditis and Sepsis (ESGBIES). Bloodstream infections - Standard and progress in pathogen diagnostics. Clin Microbiol Infect. 2020 Feb;26(2):142-150. doi: 10.1016/j.cmi.2019.11.017. Epub 2019 Nov 22. PMID 31760113
- [Background] Dubourg G, Lamy B, Ruimy R. Rapid phenotypic methods to improve the diagnosis of bacterial bloodstream infections: meeting the challenge to reduce the time to result. Clin Microbiol Infect. 2018 Sep;24(9):935-943. doi: 10.1016/j.cmi.2018.03.031. Epub 2018 Mar 29. PMID 29605563
- [Background] T Babin, T Dedole, P Bouvet, PR Marcoux, M Gougis, P Mailley (2023) Electrochemical label-free pathogen identification for bloodstream infections diagnosis: towards a machine learning based smart blood culture bottle. Sensors and Actuators B. (open access) https://doi.org/10.1016/j.snb.2023.133748